CLINICAL TRIAL: NCT02226133
Title: A Clinical Trial to Evaluate Safety and Effectiveness of the LAAx,Inc., TigerPaw System II LAA Exclusion Device for the Exclusion of the Left Atrial Appendage Via Video-Assisted Thoracoscopic Surgery ("VATS")
Brief Title: Video-Assisted Left Atrial Appendage Exclusion Trial
Acronym: VALET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped for operational reasons
Sponsor: LAAx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D&D CIP-0030
Record Dates: First submitted 2014-08-23; First posted 2014-08-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exclusion of Left Atrial Appendage (Experimental): Left Atrial Appendage (LAA) occlusion, using the LAAx, Inc. TigerPaw® System II (delivery system and implant/Fastener) using VATS techniques,
  Interventions: Device: LAAx, Inc. TigerPaw® System II

INTERVENTIONS:
Device: LAAx, Inc. TigerPaw® System II — Exclusion of Left Atrial Appendage.
  Other Names: LAAx,Inc. TigerPaw System

SUMMARY:
Exclusion of the LAA(Left Atrial Appendage) using the TigerPaw II System with VATS technique is safe and effective.

DETAILED DESCRIPTION:
The objective of this confirmatory study is to demonstrate that the LAAx, Inc. TigerPaw® II System can be safely and effectively used to exclude the Left Atrial Appendage (LAA) during cardiac surgery utilizing thoracoscopic camera and light source and thus remove, from the cleared indication for use, the direct vision limitation.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age;
2. Capable and willing to give informed consent;
3. Able and willing to complete a 30 day ± 7 day follow-up evaluation;
4. Ejection fraction ≥ 30%;
5. Life expectancy of > 1 year;
6. Stroke Risk (CHADS score of ≥ 1), CHADS scoring: CHF=1 point, Hypertension (or treated hypertension) = 1 point, Age > 75 = 1 point, Diabetes = 1 point, Prior stroke or TIA = 2 points;
7. Subjects suitable for elective Video-Assisted Thoracoscopic Surgical (VATS) procedure(s) including, but not limited to, cardiac surgery for one or more of the following:

   1. mitral valve repair or replacement,
   2. aortic valve repair or replacement,
   3. tricuspid valve repair or replacement,
   4. coronary artery bypass procedures,
   5. concomitant surgical (ablation or cut and sew) Maze procedure and other ablation procedures
   6. hybrid procedures including combination surgical and interventional procedures and surgical procedures with a combination of left and right thoracic access sites

Exclusion Criteria:

1. Previous cardiac surgery;
2. Active systemic or cutaneous infection or inflammation;
3. Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids not including intermittent use of inhaled steroids for respiratory diseases;
4. Known, significant history of bleeding diathesis, coagulopathy, von Willebrand's disease or current platelet count < 100,000 cells/mm3, baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
5. Severe co-existing morbidities having a life expectancy of less than 1 year;
6. Currently involved in any other investigational clinical trials that have not completed their primary endpoint or that may interfere with the TigerPaw study results;
7. Thrombus in the LAA/LA;
8. NYHA Class IV heart failure symptoms;
9. Mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study and to cooperate with follow-up requirements;
10. Preoperative need for an intra-aortic balloon pump;
11. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
12. Females who are pregnant, planning to become pregnant within 1 month of the procedure, or lactating;
13. Extreme morbid obesity (BMI greater than 45 kg/m2);
14. Any active medical condition that would preclude the patient from completing the study or would result in an unreasonable risk;
15. Contraindication to Transesophageal Echocardiography (TEE);
16. Need for emergent cardiac surgery (e.g., cardiogenic shock);
17. Creatinine >200 umol/L;
18. Renal failure requiring dialysis or hepatic failure;
19. A known drug and/or alcohol addiction;
20. Concurrent chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
rate of device related adverse and serious adverse events | 30 (plus or minus 7) days

SECONDARY OUTCOMES:
Exclusion of the Left Atrial Appendage | 30 days
  Primary effectiveness will be measured by the percentage of patients with exclusion of the LAA assessed intraoperatively via endoscopic image and transesophageal echocardiography (TEE).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - ValleyCare Health System-Pleasanton, Pleasanton, California
  - UMD School of Medicine, Baltimore, Maryland
  - Geisinger Heart Institute, Danville, Pennsylvania
  - Lankenau MOB East, Wynnewood, Pennsylvania